CLINICAL TRIAL: NCT00581191
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SLV-351 Administered Orally to Healthy Subjects
Brief Title: Study Evaluating the Safety and Tolerability of Single Ascending Dose (SAD) SLV-351 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 3233A1-1000
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: SAD; Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- 1 (Experimental): 0.5 mg SLV-351 (fasted)
  Interventions: Drug: SLV-351
- 2 (Experimental): 1 mg SLV-351 (fasted)
  Interventions: Drug: SLV-351
- 3 (Experimental): 2.5 mg SLV-351 (fasted)
  Interventions: Drug: SLV-351
- 4 (Experimental): 5 mg SLV-351 (fasted)
  Interventions: Drug: SLV-351
- 5 (Experimental): 10 mg SLV-351 (fasted)
  Interventions: Drug: SLV-351
- 6 (Experimental): 15 mg SLV-351 (fasted)
  Interventions: Drug: SLV-351
- 7 (Experimental): 20 mg SLV-351 (fasted)
  Interventions: Drug: SLV-351
- 8 (Experimental): 30 mg SLV-351 (fasted)
  Interventions: Drug: SLV-351
- 9 (Experimental): xx mg SLV-351 (fasted and fed)
  Interventions: Drug: SLV-351

INTERVENTIONS:
Drug: SLV-351 — SLV-351 capsules taken once

SUMMARY:
Safety and tolerability of single oral doses in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men, aged 18-50 years.
* Women of nonchildbearing potential, aged 18-50 years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Safet and tolerability | 35 days

SECONDARY OUTCOMES:
PK and PD | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer